CLINICAL TRIAL: NCT03866018
Title: Contribution of Physical Activity to Self-esteem and Motivation in Older Adults With Minor to Major Cognitive Disorders Such as Alzheimer's Disease or Related Disorders
Acronym: APAMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-AOI-01
Record Dates: First submitted 2019-02-27; First posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-02

CONDITIONS: Cognitive Disorders
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted physical activity (Experimental): Patients will participate in an adapted physical activity workshop.
  Interventions: Other: Adapted physical activity

INTERVENTIONS:
Other: Adapted physical activity — 12 sessions of one hour of adapted physical activity.

SUMMARY:
Alzheimer's disease is the leading cause of dementia in people over 60 years of age. It is characterized by a decline in memory, learning ability and other cognitive domains (language, gnosis, praxis, attention), with a gradual progression of cognitive and behavioral symptoms. Because of the difficulties it causes in carrying out daily living activities, it has a very significant impact on the autonomy of patients suffering from it.

To date, there are various non-drug strategies available to manage these difficulties. Thus, in recent years, more and more studies have shown the benefits that can be gained by several patients care including physical activity, on cognitive function and general quality of life of the elderly people without cognitive impairment but also for patients suffering from Alzheimer's disease or a related pathology.

The objective of this study is to evaluate the effectiveness of adapted physical activity on self-esteem and motivation in patients with neurocognitive disorders. Stimulation groups are proposed within the Claude Pompidou Institute. Within these groups we offer an adapted physical activity program that we have developed in our department. More specifically, it is a study that aims to evaluate the impact of physical activity on the self-esteem and motivation of patients who perform these exercises for 12 weeks, at the rate of one hour per week.

The interest of this study lies in the validation of the effectiveness of such patient care, which would make it possible to promote its dissemination and strengthen the accessibility of this type of non-drug management to elderly people suffering from neurocognitive disorders.

DETAILED DESCRIPTION:
Alzheimer's disease is the leading cause of dementia in people over 60 years of age. It is characterized by a decline in memory, learning ability and other cognitive domains (language, gnosis, praxis, attention), with a gradual progression of cognitive and behavioral symptoms. Because of the difficulties it causes in carrying out daily living activities, it has a very significant impact on the autonomy of patients suffering from it.

To date, there are various non-drug strategies available to manage these difficulties. Thus, in recent years, more and more studies have shown the benefits that can be gained by several patients care including physical activity, on cognitive function and general quality of life of the elderly people without cognitive impairment but also for patients suffering from Alzheimer's disease or a related pathology.

The objective of this study is to evaluate the effectiveness of adapted physical activity on self-esteem and motivation in patients with neurocognitive disorders. Stimulation groups are proposed within the Claude Pompidou Institute. Within these groups we offer an adapted physical activity program that we have developed in our department. More specifically, it is a study that aims to evaluate the impact of physical activity on the self-esteem and motivation of patients who perform these exercises for 12 weeks, at the rate of one hour per week.

The interest of this study lies in the validation of the effectiveness of such patient care, which would make it possible to promote its dissemination and strengthen the accessibility of this type of non-drug management to elderly people suffering from neurocognitive disorders.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ≥ 60 years old
* MMSE score between 4 and 26 / 30
* Diagnosis of minor to major NeuroCognitive Disorder of the Alzheimer type or multiple etiology;
* Subject without a major hearing or visual impairment;
* Subject not presenting any contraindications to the practice of adapted physical activity;
* Subject affiliated to Social Security System;
* Signing informed consent

Exclusion Criteria:

* < 60 years
* Medical indications: Recent or unstable cardiovascular events: ECG changes, unstable angina, uncontrolled arrhythmia, 3rd degree BAV, acute heart failure.
* MMSE score < 4
* Subject already engaged in appropriate physical activity
* Subject with a perceptual disorder (AMD, deafness...)
* Subject with a motor disability
* Subject under guardianship, curatorship or safeguard of justice
* Persons deprived of their liberty (administrative or judicial)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of patient self-esteem | At 4 months
  Rosenberg self-esteem scale
Improvement of patient motivation | At 4 months
  EAD scale
Improvement of patient apathy | At 4 months
  Apathy inventory

SECONDARY OUTCOMES:
Quantitative assessment of physical activity | At 4 months
  questionnaire for caregivers
Patient satisfaction | At 4 months
  satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Claude Pompidou - Centre Mémoire de Ressources et de Recherche du CHU de Nice, Nice, France